CLINICAL TRIAL: NCT02053662
Title: Biomarker Identification for Bladder Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: No publishable data was acquired from the study and the primary researcher left over 5 years ago.
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Arnab Chakravarti, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-12158
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bladder cancer tissue samples, blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder Cancer Patients: Patients with muscle invasive bladder cancer. A sample collection of donated cancer and normal adjacent tissues, blood and urine which will be prospectively obtained from patients through the Tissue Procurement Shared Resources (TPSR) and The Ohio State University Comprehensive Cancer Center Biospecimen and Biorepository Resource (BBR) as needed.
  Interventions: Procedure: Sample Collection

INTERVENTIONS:
Procedure: Sample Collection — A collection of donated cancer and normal adjacent tissues, blood and urine which will be prospectively obtained from patients through the Tissue Procurement Shared Resources (TPSR) and The Ohio State University Comprehensive Cancer Center Biospecimen and Biorepository Resource (BBR) as needed.

SUMMARY:
To develop a simple blood and urine test that we would perform before patients start their treatment to predict the risk that their bladder cancer might come back. To develop this test the investigators plan to analyze blood, urine and cancer tissue from bladder cancer patients and follow them closely during and after treatment. This will include looking for changes in proteins and genes that might play a role in bladder cancer biology. The investigators will then compare the information obtained from the studies of blood, urine and cancer tissue between patients that are cured and those whose cancer comes back. The knowledge about these differences between patients can then potentially be used to develop a blood or urine test to tell us who has a high risk for having bladder cancer come back.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old.
* Patients suspected, clinically diagnosed, or histologically diagnosed bladder cancer.
* Patients undergoing cystoscopy without cancer suspicion.
* Ability to give an informed consent.

Exclusion Criteria:

* Patients receiving concurrent therapy for a second malignancy.
* < 18 years old.
* Inability to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected muscle-invasive bladder cancer and appropriate control population
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Identify novel biomarkers for bladder cancer | up to 5 years
  Predict and detect bladder cancer recurrence, specifically through development of biomarkers using bladder cancer tissue samples as well as blood and urine samples. Detect the recurrence of disease through development of blood and urine biomarkers using pre-therapy and post-therapy biospecimens.

CONTACTS AND LOCATIONS:
Overall Officials: Arna Chakravarti, MD, Principal Investigator — The Ohio State University Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu